CLINICAL TRIAL: NCT04734015
Title: Family-Based, Culturally-Centered Diabetes Intervention With Ojibwe Communities
Brief Title: Together Overcoming Diabetes
Acronym: TOD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DK091250; 5R01DK091250-07 (NIH); IRB00010045 (Other: JHSPH IRB)
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Family Intervention; Lifestyle Intervention; Indigenous; American Indian; Native American
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized Waitlist Control Design. Adult/youth participant dyads will be randomized to either the intervention group or the wait-list control group after eligibility screening, enrollment and completion of the baseline assessment.
  The intervention group will receive the 6-month intervention and 6-month maintenance phase immediately; the wait-list will receive standard care for 24 months and will then receive the intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An Independent Evaluation team will conduct assessments and be blinded to participant randomization status. The investigators will also be blinded to randomization status during data collection and initial analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Together Overcoming Diabetes (TOD) curriculum (Experimental): A randomized waitlist control trial (RCT) design will be employed with 81 family dyads (adult caregiver and youth) randomly assigned to the Intervention group (Group A): Together Overcoming Diabetes (TOD).
  Group A participant dyads will be monitored via assessment of applicable biometric, psychosocial and behavioral outcomes at baseline, 3-months into intervention delivery, 6 months after baseline (post intervention), 12 months, 18 months, and 24 months.
  Interventions: Behavioral: Together Overcoming Diabetes (TOD)
- Waitlist Control (No Intervention): A randomized waitlist control trial (RCT) design will be employed with 81 family dyads (adult caregiver and youth) randomly assigned to the Waitlist Control group (Group B). Waitlist family dyads will not initially receive the intervention. They will be monitored via assessment of applicable biometric, psychosocial and behavioral outcomes at baseline, 3-months into intervention delivery, 6 months after baseline (post intervention), 12 months, 18 months, and 24 months.
  Waitlist participant dyads will begin to receive the intervention program (TOD) approximately 24 months (2 years) after enrollment in the RCT.

INTERVENTIONS:
Behavioral: Together Overcoming Diabetes (TOD) — Curriculum approaches health through a holistic lens of spiritual, mental, physical and emotional wellness. American Indian Family Health Coaches conduct motivational interviewing to help participant dyads (adult caregivers with Type 2 diabetes and their youth) set attainable goals and work through obstacles to reach those goals.
  Other Names: Niwii-shaagoojitoomin Izhi-Maamawi (we defeat/overcome it together)
  Arms: Together Overcoming Diabetes (TOD) curriculum

SUMMARY:
Together Overcoming Diabetes (TOD) is a culturally tailored, family-based type 2 diabetes management and preventive intervention.

Participants in this trial are American Indian adult caregivers diagnosed with type 2 diabetes and their youth, aged 10-16 years at enrollment. Adult/youth participant dyads will be enrolled across 5 Ojibwe tribal communities. Consenting participant dyads will be randomized into one of two groups:

Group A: begin the intervention program immediately; Group B (waitlist): begin the intervention program in 2 years.

Both groups will complete assessments with study staff at baseline, 3, 6, 12, 18, and 24 months to assess HbA1c, cholesterol, blood pressure (adults), biometric measures, and psychosocial and behavioral outcomes (adults and youth).

The 14-lesson intervention program will be delivered in the participant's home by local Family Health Coaches over a 6-month period.

Upon completion of the intervention, participants may also be invited to participate in a "Ripple Effects Mapping" (REM) session for discussions, and mapping of the intervention effects.

DETAILED DESCRIPTION:
Together Overcoming Diabetes (TOD) is a culturally tailored, family-based type 2 diabetes management and preventive intervention. The program activates family and cultural practices that encourage healthy diets and physical activities, promotes coping skills for dealing with stress, and reconnects families via a home-based intervention taught by American Indian (AI) paraprofessional Family Health Coaches.

Evaluation of TOD for this trial will happen via Community Based Participatory Research (CBPR). The study team will enroll "target" adult caregivers diagnosed with type 2 diabetes and their youth, ages 10-16 years at enrollment, with the goal of tapping motivational reciprocity between the two generations. The work involves collaboration with five Ojibwe tribal communities in the midwestern U.S. to implement a randomized controlled study with a wait-list design respectful of cultural norms of inclusion.

The study will evaluate effectiveness of the intervention on adult physiological (primary outcome = HbA1c), behavioral, and mental health and children's psychosocial, familial, behavioral and physiological risk and protective factors for diabetes. The research will also identify stress-coping mechanisms that mediate the impact of the intervention on health. A novel collaborative, qualitative evaluation technique will map potential "ripple effects" of the intervention within families and communities. If effective, the intervention will promote dissemination and scaling with tribal health coaches, community involvement, and stakeholder (health providers, health and human service agencies) input.

ELIGIBILITY:
Inclusion Criteria:

ADULT (target participants)

* Are greater than 18 years of age
* Self-identify as American Indian
* Have a completed verification form from a healthcare provider indicating a confirmed diagnosis of type 2 diabetes
* Live on or within 30 miles of participating reservations
* Are a caregiver to a 10-16 year-old who lives in their home
* Are willing to be randomly put into Group A (intervention) or Group B (waitlist control)
* Are willing to complete all lessons and assessments
* Speak and read English
* Are not cognitively or visually impaired (able to review and sign informed consent and complete assessments)

YOUTH

* 10 -16 years of age
* Self-identify as American Indian
* Live with an adult who has joined the study
* Are willing to be randomly put into Group A or Group B
* Are willing to complete all lessons and assessments
* Speak and read English
* Are not cognitively or visually impaired (able to review and sign informed consent and complete assessments)

Exclusion Criteria:

ADULTS (target participants)

* Are not American Indian
* No confirmed type 2 diabetes diagnosis
* Not a caregiver to a youth ages 10-16 in their home
* Does not live within the distance inclusion criteria
* Is unable to complete the study procedures
* Has comorbidity(ies) that may have an impact on type 2 diabetes management

YOUTH

* Are not American Indian
* Do not fall within the specified age range of 10-16 years at time of enrollment
* Do not have an enrolled Adult caregiver
* Unable to read and speak English
* Not willing to complete the study procedures

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Adult Participant Fasting HbA1c | Day 0, Month 3, Month 6, Month 12, Month 18, and Month 24
  Change in hemoglobin A1c

SECONDARY OUTCOMES:
Change in BMI/zBMI - Adult and Youth participants | Day 0, Month 3, Month 6, Month 12, Month 18, and Month 24
  zBMI change as indication of weight loss
Change in Depression and Depressive symptoms - Adult and Youth participants | Day 0, Month 3, Month 6, Month 12, Month 18, and Month 24
  Patient Health Questionnaire (PHQ-9) Adult and Adolescent versions. Scoring ranges from 0 to 3. Higher total score equates to worse outcome.

OTHER OUTCOMES:
Change in Physical Activity - Adult and Youth participants | Day 0, Month 6, Month 12, and Month 24
  Survey questions will ask about physical activity duration, frequency, intensity. Higher score equates to better outcome.
Change in Communal Mastery - Adult and Youth participants | Day 0, Month 6, Month 12, and Month 24
  Communal Mastery as a Coping Resource. Scoring ranges from 0 to 3. Higher score equates to better outcome.
Change in Diabetes Empowerment - Adult participants | Day 0, Month 6, Month 12, and Month 24
  Diabetes Empowerment Scale (short form, Anderson, et al., 2003). Scoring ranges from 0 to 3. Higher score equates to better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Walls, PhD, Principal Investigator — Johns Hopkins University, Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University Great Lakes Hub, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walls ML, Sittner KJ, Gomez GJ, Cole RE, Perkins SR, Steinberg RI, Forsberg AK, Haroz EE, Barlow A. Trial and Participant Characteristics of a Home-Visiting Diabetes Intervention: The Together Overcoming Diabetes Study. J Diabetes Res. 2025 Apr 24;2025:6591307. doi: 10.1155/jdr/6591307. eCollection 2025. PMID 40313359